CLINICAL TRIAL: NCT04894799
Title: Effects of Vestibular Stimulation and Neurodevelopmental Technique on Hypotonic Cerebral Palsy While Controlling the Gender
Brief Title: Vestibular Stimulation and Neurodevelopmental Technique on Hypotonic Cerebral Palsy While Controlling the Gender
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00983 Sadaf Zahra
Record Dates: First submitted 2021-05-19; First posted 2021-05-20 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Cerebral Palsy; Hypotonia
Keywords: developmental milestones; hypotonia; vestibular stimulation
MeSH Terms: conditions — Cerebral Palsy; Muscle Hypotonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular stimulation (Experimental): all participants will be given Infant Swing activity for one hour, trice a day for first 4 weeks. After that, in 5th and 6th weeks, all participants will be given Infant Swing for 30 minutes and frog swing for 30 minutes for two weeks. Next 7th and 8th weeks, Infant Swing (30 minutes) and prone on frog swing feet touching the floor (30 minutes), trice a day will be applied. In 9th week, Infant swing and normal playground swing for 30,30 minutes will be given to all participants, trice a day. In Last week of intervention i.e., 10th week, all participants will be given Infant Swing for 30 minutes and standing on platform swing (30 minutes) trice a day.
  Interventions: Other: Vestibular stimulation
- Neck Control facilitation exercises (Active Comparator): all participants will be given Neck Control facilitation exercises using Bobath Approach of low tone facilitation method, for one hour, trice a day for first 4 weeks. After that, in 5th and 6th weeks, all participants will be given Neck Control facilitation exercises for 30 minutes and sitting facilitation Exercises with trunk weight shifting for 30 minutes, trice a day. Next 7th and 8th weeks, Neck Control facilitation exercises (30 minutes) and sitting facilitation exercises with trunk weight shifting and kneeling weight bearing (30 minutes), trice a day will be applied. In 9th and 10th weeks, Neck Control facilitation exercises, sitting and kneeling weight bearing and standing with trunk elongation will be given to all participants for one hour, trice a day.
  Interventions: Other: Neck Control facilitation exercises

INTERVENTIONS:
Other: Vestibular stimulation — In Vestibular Stimulation (VS) group, all participants will be given Infant Swing activity for one hour, trice a day for first 4 weeks. After that, in 5th and 6th weeks, all participants will be given Infant Swing for 30 minutes and frog swing for 30 minutes for two weeks. Next 7th and 8th weeks, Infant Swing (30 minutes) and prone on frog swing feet touching the floor (30 minutes), trice a day will be applied. In 9th week, Infant swing and normal playground swing for 30,30 minutes will be given to all participants, trice a day. In Last week of intervention i.e., 10th week, all participants will be given Infant Swing for 30 minutes and standing on platform swing (30 minutes) trice a day.
  Arms: Vestibular stimulation
Other: Neck Control facilitation exercises — all participants will be given Neck Control facilitation exercises using Bobath Approach of low tone facilitation method, for one hour, trice a day for first 4 weeks. After that, in 5th and 6th weeks, all participants will be given Neck Control facilitation exercises for 30 minutes and sitting facilitation Exercises with trunk weight shifting for 30 minutes, trice a day. Next 7th and 8th weeks, Neck Control facilitation exercises (30 minutes) and sitting facilitation exercises with trunk weight shifting and kneeling weight bearing (30 minutes), trice a day will be applied. In 9th and 10th weeks, Neck Control facilitation exercises, sitting and kneeling weight bearing and standing with trunk elongation will be given to all participants for one hour, trice a day.
  Arms: Neck Control facilitation exercises

SUMMARY:
there is no such article found who specifies the effects of sensory integration therapies like vestibular stimulation technique or developmental milestone while controlling the gender of children with cerebral palsy. So, there is a need to do more research work on this in future to find out best treatment approach for children with cerebral palsy of their respective gender. That is why this study will focus on the results of vestibular stimulation and neurodevelopmental technique while controlling the Gender distribution of both intervention groups to find out the effects of these interventions that wither, they have some influence on the participants or not.

DETAILED DESCRIPTION:
Bobath concept of neurodevelopment in children with cerebral palsy, is a problem-solving approach to the assessment and treatment of individuals with disturbances of tone, movement, and function due to a lesion of CNS, the goal of treatment is to optimize function by improving postural control and selective movement through facilitation. But also, no study found which specifically focuses the improvements on boys and girl's ratio or their gender-based improvements of tone or developmental milestones.

Different swings such as Infant Swing, frog swing, platform swing will be included as mode of Vestibular stimulation treatment. On the other side, Stimulation of vestibular system improved child's postural control and motor function in many studies.

ELIGIBILITY:
Inclusion Criteria:

* Hypotonic CP
* GMFM-88 ranges: With true score of zero (0) = does not initiates i.e., head control absent at age of 6 months
* Tone: 6 months infants total scoring ≤ 54 and 8 month or more total scoring ≤ 68 on Infant Neurological international Battery Scoring Sheet will be included.

Exclusion Criteria:

* Children with other Abnormalities and pathologies like Down syndrome, Joubert Syndrome

  * Children Undergone any kind of surgery like reconstruction surgeries for congenital defects of eyes, head, neck or all four limbs of the body
  * Children with other type of Cerebral Palsy (CP) like Spastic (Hypertonic), Choreoathetoid, Dystonic, Ataxia, Athetoid and mixed CP
  * Children with any other neurological deficits, Mentally Challenged.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Self representation of gender identity
Enrollment: 24 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Infant Neurological International Battery | 10 weeks
  Infant Neurological International Battery ( INFANIB) is the developmental screening tool used for the assessment of neuromotor development in neonates and infants aged 1-18 months. The score of each item is mentioned in the score sheet itself based upon age and calculating total score will determine the neuromotor state of infants.
GMFM-88 | 10 weeks
  It is a Standardized Observational Instrument designed and validated to measure change in gross motor function over time in children with Cerebral Palsy. The GMFM-88 item scores can be summed to calculate raw and percent scores for each of the five GMFM dimensions of interest, selected goal areas and a total GMFM-88 score.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, Principal Investigator — Riphah International University
Locations (1):
- Helping Hand Comprehensive Rehabilitation Center, Chakwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No